CLINICAL TRIAL: NCT04225026
Title: A Phase 2a Open-Label Trial of the Effects of Intravenous GC4419 on the Incidence and Severity of Esophagitis in Subjects Receiving Chemoradiotherapy for Lung Cancer
Brief Title: Effects of Intravenous GC4419 on the Incidence and Severity of Esophagitis Due to Chemoradiotherapy for Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of study enrollment
Sponsor: Galera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTI-4419-203
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Results first posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2022-06

CONDITIONS: Esophagitis
MeSH Terms: conditions — Esophagitis | interventions — avasopasem manganese

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GC4419 (avasopasem manganese) (Experimental)
  Interventions: Drug: GC4419 (avasopasem manganese)

INTERVENTIONS:
Drug: GC4419 (avasopasem manganese) — 90 mg, by 60-minute IV infusion, prior to each fraction of RT
  Other Names: Avasopasem manganese

SUMMARY:
GTI-4419-203 will be an open-label, multi-center study to evaluate GC4419 (avasopasem manganese) administered intravenous (IV) for the reduction of radiation induced esophagitis in subjects receiving chemoradiotherapy for unresectable Stage 3A/3B or post-operative Stage 2B Non-Small Cell Lung Cancer (NSCLC) or Small Cell Lung Cancer (SCLC) treatable with chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects scheduled to be treated with (definitive or adjuvant) radiation therapy in combination with chemotherapy once daily for Stage 3A/3B or post-operative Stage 2B NSCLC or limited stage SCLC
2. Treatment plan for subjects show that 5 cm of the esophagus for at least one surface, is included in the 60 Gy isodose volume. Dose volume histograms show esophagus dose exposure meet V38>30% and/or V60>20%
3. Age 18 years or older
4. ECOG performance status ≤ 2
5. Adequate hematologic, renal and liver function
6. Use of highly effective contraception

Exclusion Criteria:

1. Metastatic disease
2. Prior radiation therapy to the region of the study cancer
3. Subjects not receiving chemotherapy
4. Grade 2 or greater esophagitis at baseline
5. Inability to provide information in the electronic symptom-reporting device
6. Receiving any approved or investigational immunotherapy, targeted therapy, hormone therapy, or biologic therapy
7. Participation in another clinical trial or use of another investigational agent within 30 days of first does of GC4419
8. Malignant tumors other than the current lung cancer within the last 5 years
9. Previous diagnosis of pneumonitis
10. Untreated, active infectious disease requiring systemic anti-infective therapy
11. Untreated HIV or active hepatitis B/C
12. Females who are pregnant or breastfeeding
13. Known allergies or intolerance to chemotherapy and similar platinum-containing compounds
14. Requirement for concurrent treatment with nitrates or other drugs that may create a risk for a precipitous decrease in blood pressure
15. Clinically significant heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2022-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Kennedy, MD, Study Chair — Chief Medical Officer
Locations (12):
- United States (12):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Tampa General Hospital, Tampa, Florida
  - IACT Health, Columbus, Georgia
  - University of Iowa, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - Cancer Care St. Joseph/Mosaic Life Care, Saint Joseph, Missouri
  - Hackensack Meridian Health, Montclair, New Jersey
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - St. Francis Hospital, Greenville, South Carolina
  - Spartanburg Regional Medical Center - Gibbs Cancer Center, Spartanburg, South Carolina
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Providence Regional Cancer Partnership, Everett, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- GC4419: GC4419: 90 mg, by 60-minute IV infusion, prior to each fraction of RT
Period: Overall Study
Arm/Group | GC4419
Started (Safety analysis Population: This population included all subjects who received at least 1 dose of study medication.) | 39
Primary Efficacy Population | 35 (The Primary Efficacy Population includes all subjects who received at least one dose of GC4419 and either a.)completed their radiation therapy course of treatment or b.)discontinued their radiation therapy course of treatment but are known to have had acute radiation esophagitis.)
Per Protocol Population (The Per Protocol Population included those subjects that completed chemoradiotherapy and at least 5 weeks of GC4419) | 29
Completed | 15
Not Completed | 24
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 1
Not completed — Other | 1
Not completed — Death | 11
Not completed — Study Terminated Early By Sponsor | 7

BASELINE CHARACTERISTICS:
Population: The primary efficacy population includes all subjects who received at least one dose of GC4419 and either a.) completed their radiation therapy course of treatment or b.) discontinued their radiation therapy course of treatment but are known to have had acute radiation esophagitis.
Arm/Group | GC4419
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: There were 39 subjects enrolled to the study but only 35 subjects were included in the primary efficacy analysis population based on the primary efficacy population definition.
  years | 65.1 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Their were 39 subjects enrolled to the study but only 35 subjects were included in the analysis population based on the primary efficacy population definition.
  Participants
    Female | 17
    Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Their were 39 subjects enrolled to the study but only 35 subjects were included in the analysis population based on the primary efficacy population definition.
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 38
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Their were 39 subjects enrolled to the study but only 35 subjects were included in the analysis population based on the primary efficacy population definition.
  Participants
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 2
    White | 36
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Population: Their were 39 subjects enrolled to the study but only 35 subjects were included in the analysis population based on the primary efficacy population definition.
  participants
    United States | 39
Type of Lung Cancer [Number; unit: participants] — Population: Their were 39 subjects enrolled to the study but only 35 subjects were included in the analysis population based on the primary efficacy population definition.
  participants
    NSCLC | 32
    SCLC | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With of Acute Radiation Esophagitis (Defined as Grade >/= 2; NCI CTCAE Version 5) Through the End of Chemoradiotherapy for Non-Small Cell Lung (NSCLC) or Small Cell Lung Cancer (SCLC) When Avasopasem Was Added.
Description: Those subjects in the primary efficacy population that experience acute radiation esophagitis (Grade >/=2; NCI CTCAE version 5) through the end of chemoradiotherapy for NSCLC or SCLC when treated with avasopasem.
  NCI CTCAE Grading:
  Grade 1: asymptomatic; clinical or diagnostic observations only; intervention not indicated Grade 2: symptomatic; altered eating/swallowing; oral supplements indicated Grade 3: severely altered eating/swallowing; tube feeding, total parental nutrition (TPN) or hospitalization Grade 4: life-threatening consequences; urgent operative intervention indicated Grade 5: death
Time Frame: From the first radiation therapy fraction through the end of the study treatment period, which is estimated to be 6 weeks.
Population: Primary Efficacy Population included all subjects who received at lease 1 dose of GC4419 (avasopasem manganese) and either completed their radiation therapy or discontinued their radiation therapy early but were known to have had acute radiation esophagitis.
Measure: Count of Participants; unit: Participants
Arm/Group | GC4419 (Avasopasem Manganese)
Number analyzed (Participants) | 32
Participants
  Condition Not Present | 7
  Grade 1 | 6
  Grade 2 | 17
  Grade 3 | 2
  Grade 4 | 0
  Grade 5 | 0

2. Secondary Outcome: Number of Subjects With of Acute Radiation Esophagitis (Defined as Grade >/= 2; NCI CTCAE Version 5) Through 4 Weeks After Completion of Chemoradiotherapy
Description: Those subjects in the in the primary efficacy population that experience Grade >/= 2 (NCI CTCAE version 5) acute radiation esophagitis through 4 weeks after completion of chemoradiotherapy for NSCLC or SCLC when treated with avasopasem.
  NCI CTCAE Grading:
  Grade 1: asymptomatic; clinical or diagnostic observations only; intervention not indicated Grade 2: symptomatic; altered eating/swallowing; oral supplements indicated Grade 3: severely altered eating/swallowing; tube feeding, total parental nutrition (TPN) or hospitalization Grade 4: life-threatening consequences; urgent operative intervention indicated Grade 5: death
Time Frame: From the first radiation therapy fraction through 4 weeks after the completion of chemoradiotherapy, which is estimated to be 10 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GC4419
Number analyzed (Participants) | 34
Participants
  Condition Not Present | 19
  Grade 1 | 4
  Grade 2 | 10
  Grade 3 | 1
  Grade 4 | 0
  Grade 5 | 0

3. Secondary Outcome: Number of Subjects With Acute Severe Radiation Esophagitis (Defined as Grade 3-4; NCI CTCAE Version 5) Through Completion of Chemoradiotherapy.
Description: Those subjects in the per protocol population that experienced Grade 3-4 acute radiation esophagitis through the completion of chemoradiotherapy.
  NCI CTCAE Grading:
  Grade 1: asymptomatic; clinical or diagnostic observations only; intervention not indicated; Grade 2: symptomatic; altered eating/swallowing; oral supplements indicated; Grade 3: severely altered eating/swallowing; tube feeding, total parental nutrition (TPN) or hospitalization; Grade 4: life-threatening consequences; urgent operative intervention indicated; Grade 5: Death.
Time Frame: From the first radiation therapy fraction through the completion of chemoradiotherapy, which is estimated to be 6 weeks.
Population: Per protocol population defined as those subjects completing chemoradiation therapy and at least 5 weeks of GC4419
Measure: Count of Participants; unit: Participants
Arm/Group | GC4419 (Avasopasem Manganese)
Number analyzed (Participants) | 29
Participants
  Condition Not Present | 7
  Grade 1 | 6
  Grade 2 | 13
  Grade 3 | 1
  Grade 4 | 0
  Grade 5 | 0
  Assessment Not Performed | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline (Study Day 1) until 30 days post the last day of radiation therapy (approximately 10 weeks).
Arm/Group | GC4419
All-Cause Mortality (participants affected / at risk) | 11/39
Serious Adverse Events (participants affected / at risk) | 15/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GC4419 (N=39)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Adult Failure to Thrive (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Corona Virus Infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Non Cardiac Chest Pain (General disorders) | 2 (2)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Atrial Tachycardia (Cardiac disorders) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Confusional State (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GC4419 (N=39)
Paraesthesia (Nervous system disorders) | 8 (84)
Nausea (Gastrointestinal disorders) | 22 (60)
Dysphagia (Gastrointestinal disorders) | 20 (53)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 11 (33)
Fatigue (General disorders) | 24 (32)
Vomiting (Gastrointestinal disorders) | 15 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution shall provide Sponsor with an advance copy of any proposed publication at least 45 days prior to the planned date of submission or presentation and Sponsor shall have 45 days to review. Institution may be asked by Sponsor to delete confidential information, consider reasonable changes requested by Sponsor or delay proposed submission for additional period, not to exceed 90 days, to protect the potential patentability of any technology.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/26/NCT04225026/Prot_SAP_000.pdf